CLINICAL TRIAL: NCT06950112
Title: Comparison Between Individualized PEEP Ventilation Guided by Driving Pressure and Conventional Lung Protective Strategy in Obese Patients Undergoing Laparoscopic Bariatric Surgery: a Prospective Randomized Controlled Trial
Brief Title: Comparison Between Individualized PEEP Ventilation Guided by Driving Pressure and Conventional Lung Protective Strategy in Obese Patients Undergoing Laparoscopic Bariatric Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahmoud Gamal Ahmed Arakeeb (Other)
Responsible Party: Sponsor-Investigator, Mahmoud Gamal Ahmed Arakeeb, Assistant lecturer of anesthesia faculity of medicine tanta university, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 36265MD302/11/24
Record Dates: First submitted 2025-03-23; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Obese Patients With Bariatric Surgery; Lung Ultrasound Score

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group D (Driving pressure) (Experimental): Patients will be ventilated with driving pressure-guided ventilation with VT 6-8 ml /kg of predicted body weight, and after recruitment, we will return to the baseline PEEP 5 cmH2O that will be increased by 2 cmH2O until reaching the lowest possible driving pressure for every patient. Each PEEP level will be maintained for ten respiratory cycles and DP will be calculated at the last cycle.
  Interventions: Device: lung ultrasound
- Group L (Lung protective strategy) (Experimental): Patients will be ventilated with protective lung strategy with VT 6-8 ml /kg of predicted body weight, after recruitment we will return to PEEP of 8-10 cm H2O that will be maintained until the end of surgery.
  Interventions: Device: lung ultrasound
- Group P (Physiological PEEP) (Experimental): Patients will be ventilated with VT 6-8 ml /kg of predicted body weight, after recruitment we will return to physiological PEEP of 5 cm H2O that will be maintained until the end of surgery.
  Interventions: Device: lung ultrasound

INTERVENTIONS:
Device: lung ultrasound — The lung ultrasound score between 0 and 3 (0 = normal A lines, 1 = multiple separated B lines, 2 = coalescing B lines or light beam, 3 = consolidation). The aeration score will be built by the sum of the scores of the 12 segments, with a minimum of 0 and a maximum of 36 according to the aeration loss.

SUMMARY:
this study to compare the ventilation in obese patients either using Driving pressure ventilation technique or conventional protective lung strategy all by using Lung ultrasound score

ELIGIBILITY:
Inclusion Criteria:

1. patients who have a BMI 30-40 kg/m2
2. American Society of Anesthesiologists (ASA) physical status II or III
3. patients aged between 18 and 60 years,
4. patients scheduled to undergo laparoscopic bariatric surgeries.

Exclusion Criteria:

1. patients' refusal to participate in the study,
2. previous history of thoracic surgery,
3. Patients with a history of chest disease (COPD, emphysema, or pneumothorax),
4. Patients with abnormal pre-operative chest radiographs, such as pneumonia and pleural effusion,
5. Patients with right-side heart failure or impending failure,
6. Patients with known hypovolemia, and Patients with increased intracranial pressure.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
The change in lung ultrasound score | Periprocedural
  The primary outcome will be the change in Lung Ultra Sound Score between 0 and 3 (0 = normal A lines, 1 = multiple separated B lines, 2 = coalescing B lines or light beam, 3 = consolidation) from the base line.

SECONDARY OUTCOMES:
Lung compliance | Periprocedural
  Lung compliance is a measure of the expansion of the lung.
Hemodynamic parameter as oxygen saturation | Periprocedural
Hemodynamic parameter as Heart rate | Periprocedural
Hemodynamic parameter as Mean arterial blood pressure | Periprocedural
End-tidal carbon dioxide (ETCO2) | Periprocedural
Plateau Pressure (Pplat) | Periprocedural
Peak airway pressure (Ppeak) | Periprocedural
Incidence of early postoperative pulmonary complications | At the end of the surgery up to 24 hours after surgery
Length of post anesthesia care unit "PACU" stay. | At the end of the surgery up to 2 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta university, Tanta, El Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year
Access Criteria: The data will be available upon a reasonable request from the corresponding author